CLINICAL TRIAL: NCT01193712
Title: Non-Responders in Cardiac Resynchronization Therapy
Brief Title: Endocardial Pacing in On-table Non-responders in Cardiac Resynchronization Therapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: too limited number of eligible patients
Sponsor: Catharina Ziekenhuis Eindhoven (Other)
Responsible Party: Principal Investigator, Patrick Houthuizen, Patrick Houthuizen, Catharina Ziekenhuis Eindhoven
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NL26963.060.09
Record Dates: First submitted 2010-08-25; First posted 2010-09-02 (Estimated); Last update posted 2015-02-03 (Estimated); Status verified 2015-02

CONDITIONS: Heart Failure
Keywords: Electrophysiologic Techniques, Cardiac
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- on-table non-responder (Other): patients who do not show an improvement of more than or equal to 15% in LV dP/dtmax measured immediately after implantation of a cardiac resynchronization therapy device
  Interventions: Procedure: temporary left ventricular endocardial pacing
- on-table responders (No Intervention): patients who do show an improvement of more than or equal to 15% in LV dP/dtmax measured immediately after implantation of a cardiac resynchronization therapy device

INTERVENTIONS:
Procedure: temporary left ventricular endocardial pacing — a temporary pacemaker lead will be introduced through the aortic valve to evaluate the effect of left ventricular endocardial pacing. Four different pacing sites (basal and apical septal, basal and apical lateral) will be investigated with measurement of LV dP/dtmax. Afterwards, the endocardial pacing lead will be removed.
  Arms: on-table non-responder

SUMMARY:
The purpose of this study is to determine whether left ventricular endocardial pacing exhibits a greater acute hemodynamic response during biventricular pacing in patients who do not show this response to standard cardiac resynchronization therapy.

DETAILED DESCRIPTION:
Cardiac resynchronisation therapy (CRT) with biventricular pacemakers and implantable cardiac defibrillators (ICD) has proven to be a valuable therapy in selected patients with systolic heart failure, ameliorating both morbidity and mortality. However, with current selection criteria and implant technique, about 20 to 30 % of patients remain non-responders. Non-responders might be due to failing selection criteria or methodology in casu echocardiography. However, an important number of non-responders may result of sub-optimal positioning of the left ventricular lead, remote from the site of delayed activation. Endocardial left ventricular stimulation may ameliorate the shortcomings of epicardial stimulation. The advantage of an endocardial approach is the absence of phrenic nerve stimulation which regularly complicates epicardial pacing, a more predictable pacing threshold and much less restriction to position the lead in the area of interest. Transseptal left ventricular endocardial pacing has already been used in patients in whom standard epicardial pacing was not applicable.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18y
2. LVEF ≤35%
3. QRS-duration ≥0.12 seconds
4. NYHA functional class III or IV despite optimal medical therapy defined as use of angiotensin-converting enzyme inhibitors or angiotensin-II receptor blocker and beta-blockers unless they are not tolerated or contra-indicated
5. sinus rhythm or atrial fibrillation

Exclusion Criteria:

1. episode of acute heart failure ≤3 months
2. change in dosage of beta-blockers, angiotensin-converting enzyme inhibitors or angiotensin-II receptor blockers ≤3 months
3. unstable angina pectoris, acute myocardial infarction, percutaneous intervention or coronary bypass surgery ≤3 months
4. chronic atrial arrhythmias other than atrial fibrillation
5. any mechanical or biological valve prosthesis
6. atrial septal defect
7. right-to-left shunt
8. severe pulmonary hypertension (systolic pulmonary artery pressure >90 mmHg)
9. uncontrolled arterial hypertension
10. known allergy to sulphur hexafluoride
11. end-stage renal or hepatic disease
12. inability to provide written informed consent
13. pregnancy or childbearing potential without use of birth-control measurements
14. general contra-indications to magnetic resonance imaging

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-08; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
change in acute hemodynamic response to CRT defined as an increase in LV dP/dtmax of ≥10% during left endocardial pacing compared to left epicardial pacing. | baseline and 3 months

SECONDARY OUTCOMES:
improvement in NYHA functional class ≥1 | baseline and 3 months
decrease in MLWHFQ of ≥9 points | baseline and 3 months
decrease in LVESV of ≥15% | baseline and 3 months
increase in LVEF of ≥5% | baseline and 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Houthuizen, MD, Principal Investigator — Catharina Ziekenhuis Eindhoven
Locations (1):
- Catharina Ziekenhuis, Eindhoven, Netherlands